CLINICAL TRIAL: NCT06799507
Title: The Effect of Mindfulness-Based Lifestyle Support Program on Quality of Life, Lifestyle, Mindfulness Level and Treatment Outcomes in Infertile Women
Brief Title: The Effect of Mindfulness-Based Lifestyle Support Program on Infertile Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Figen Yanık, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DEU-HF-FY-01
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Fertility Disorders; Infertility (IVF Patients)
Keywords: Infertility; Mindfulness; Quality of Life; Life Style
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention: Intervention Based on Mindfulness
  Interventions: Behavioral: Interventions Based on Mindfulness
- Control (Active Comparator): Control: Routine clinical procedure
  Interventions: Other: Routine clinical procedure

INTERVENTIONS:
Behavioral: Interventions Based on Mindfulness — Affirmation, Relaxation, Mindfulness, Meditation, Healthy Lifestyle, Quality Life
  Arms: Intervention
Other: Routine clinical procedure — Routine clinical procedure
  Arms: Control

SUMMARY:
This randomized controlled trial aimed to determine whether a mindfulness-based lifestyle support program would improve quality of life, lifestyle, mindfulness, attention and meditation level and treatment outcomes in women undergoing IVF treatment.

DETAILED DESCRIPTION:
Having a diagnosis of infertility is often perceived by individuals as a physically and psychologically challenging experience. At every step of infertility treatment, women face different levels of anxiety and stress. In this direction, recent studies have emphasized the importance of acquiring fertility-supportive lifestyle behaviors, especially to eliminate infertility risk factors. It is stated that positive changes in lifestyle behaviors can positively affect treatment outcomes and quality of life. Recently, awareness-based interventions to support psychological well-being and healthy life behaviors in couples undergoing fertility treatment have gained importance in the literature. There are many psychosocial variables that can affect individuals' perception of quality of life in coping strategies of psychological interventions such as mindfulness. The reason for this is the acquisition of coping skills with more use of mindfulness skills. With the mindfulness approach, infertile women are encouraged to be open to encountering painful situations in the treatment process at any time, not to approach their pain judgmentally, and to see their experiences in the treatment process as a part of humanity. As a result, quality of life can improve by being aware of their body, emotions and thoughts.

The quality of life and lifestyle habits of women receiving fertility support are generally not a factor that is highly evaluated by health professionals. Clinical practice focuses more on medical procedures. However, in addition to medical care, psychological interventions that can support success should also be included in this treatment. Providing healthy lifestyle changes that can reduce stress and increase fertility and support fertility is very useful and necessary for public health.

It is thought that the "Mindfulness-Based Lifestyle Support Program" developed by the researchers and prepared in accordance with adult education principles will be effective in regulating the psychological well-being, quality of life and lifestyle of women receiving in vitro fertilization treatment with fertility-supportive lifestyle trainings and mindfulness practices, and will be effective in achieving more successful treatment results by positively affecting reproductive organs and hormonal balance. In addition, in order to see the effects of this mindfulness-based program more quantitatively, it is planned to follow up the women with wearable technology that gives subjective feedback on brain activities, attention and meditation levels.

The aim of this study is to evaluate the quality of life, lifestyle, mindfulness, attention and meditation levels and treatment outcomes of women receiving in vitro fertilization treatment with fertility-supportive lifestyle education in the "Mindfulness-Based Lifestyle Support Program", which was developed by the researchers as a hybrid and prepared in accordance with adult education principles, in a randomized controlled trial.

The research will be conducted as "hybrid education" face-to-face and online via zoom platform with women who apply to a university hospital IVF Center in Izmir for in vitro fertilization treatment and meet the sampling criteria reached by the researcher. In the study, infertile women will be randomized and divided into 2 groups as intervention and control. The intervention group will receive Mindfulness-based lifestyle support program, while the control group will not be subjected to any training and will receive routine clinical care. The effects of the Mindfulness-based lifestyle support program on infertile women's quality of life, lifestyle, mindfulness level, and treatment outcomes will be evaluated with scales and prepared forms, and the level of attention and meditation will be evaluated with the NeuroSky Mindwave device.

ELIGIBILITY:
Inclusion Criteria:

* Primary infertility,
* Going to undergo IVF treatment,
* Under 45 years of age,
* Having a smart phone or computer

Exclusion Criteria:

* Participate in any program related to mindfulness
* Prior mindfulness training
* Knowing/doing mindfulness practices beforehand
* Having any psychiatric disorder
* Having any chronic disease
* Disability (hearing/vision etc.)
* Attending less than 80% of the trainings (missing more than 2 Mindfulness trainings)
* Conception during research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
The Fertility Quality of Life | through study completion, average 28 days
  Fertility quality of life tool (FertiQoL): This scale is a self-rating questionnaire specifically designed to assess the quality of life of infertile patients. It has good reliability and efficacy in many countries. The Cronbach's α value of the Turkish version of FertiQoL is 0.905. The FertiQoL scale includes two modules: The Core FertiQoL module and the optional Treatment FertiQoL module. The Core FertiQoL module is divided into four domains: emotional (6 items), mind-body (6 items), relationship (6 items) and social (6 items). The optional Treatment FertiQoL module is divided into two domains: environment (6 items) and tolerability of infertility treatment (4 items). Each item has a score of 0-4 points and the total scale and subscale scores can be converted into 0-100 point scales. The higher the scores obtained from the scale, the higher the fertility-related quality of life.
Fertility Healthy Lifestyle | through study completion, average 28 days
  Fertility Healthy Lifestyle Assessment Scale (FHLAS): This is a 46-item scale developed by Bilgiç et al. to assess healthy lifestyles that contribute to improving fertility in women and men. It consists of seven sub-dimensions and is a 5-point Likert-type scale (1-strongly disagree, 2- disagree, 3 undecided, 4- agree, and 5-strongly agree). The seven sub-dimensions of the scale are emotional well-being, physical activity, sleep, nutrition, technology, hygiene and spirituality. Cronbach's Alpha value of the scale was found to be 0.87. The lowest score obtained from the scale is 46 and the highest score is 230. High scores obtained from the total scale and its sub-dimensions indicate that individuals have a lifestyle associated with healthier fertility.

SECONDARY OUTCOMES:
Mindfulness | through study completion, average 28 days
  Mindful Attention Awareness Scale (MAAS): aims to determine the general tendency to be aware of and attentive to momentary experiences in daily life. The 6-point Likert-type scale consists of 15 items and one dimension. As a result of the reliability analysis, the Cronbach Alpha internal consistency coefficient of the scale was calculated as .80 and the test-retest correlation was calculated as .86. High scores on the scale indicate high levels of mindfulness.
Attention and Meditation Level | through study completion, average 28 days
  NeuroSky Mindwave: The device will be implemented by the researcher. This wearable EEG device was developed as a direct biosensor to detect attention and meditation states by reading the electrical activity of the brain. The device features dry active technology, without the need for gel. The two metal parts of the ear clip are attached in contact with the earlobe and the sensor part is adjusted to contact the forehead above the left eye. With the help of the sensors, Attention and Meditation levels of the brain can be calculated. Measurement of the level of Mindfulness and Meditation will be obtained for both the intervention and the control group. In order to obtain a healthy signal with the device, there should be no elements such as hair, dead skin or makeup to prevent contact.
Treatment Outcome-Number of Embryos | through study completion, average 28 day
  The number of embryos, which is one of the treatment outcomes of women who completed the Mindfulness-Based Lifestyle Support Program, will be recorded in the "Treatment Outcome Form" created by the researchers. The information in the relevant form will be recorded by the researcher after the oocyte retrieval process by interviewing the women and looking at the system records.
Treatment Outcome-Pregnancy Rate | after study completion, average 10-12 day
  The pregnancy rate, which is one of the treatment outcomes of women who completed the Mindfulness-Based Lifestyle Support Program, will be recorded on the "Treatment Outcome Form" created by the researchers. The information in the relevant form will be recorded by the researcher by interviewing the women and checking the system records after the pregnancy test procedure performed approximately 10-12 days after the embryo transfer procedure.
Education Program Satisfaction | through study completion, average 28 days
  The satisfaction of the women who completed the Mindfulness-Based Lifestyle Support Program will be evaluated by the researchers by asking the women about their satisfaction with this program. It will be evaluated with a visual satisfaction scale created by the researcher, which includes a rating from 0 to 10 (0-not satisfied at all, 10-very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No